CLINICAL TRIAL: NCT04042064
Title: To Investigate the Influence of Surgery and Anesthesia on Elderly Population by Using the Comprehensive Geriatric Assessment
Acronym: CGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900881B0
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-07

CONDITIONS: Surgery and Anesthesia on Elderly; Comprehensive Geriatric Assessment; Aged
Keywords: CGA; Anesthesia for the elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhalation: Patient anesthetised with Inhalation anesthetic agents.
- TIVA (total intravenous anesthesia): Patient anesthetised with total total intravenous anesthesia.

SUMMARY:
Aging is a universal and progressive physiological phenomenon clinically characterized by degenerative changes in both the structure and the functional capacity of organs and tissues. A comprehensive geriatric assessment (CGA) has now become a standard assessment for caring for the elderly. CGA is a multidisciplinary team with the goal of improving the overall well-being of the elderly. It encompasses screening, diagnosis and treatment of the elderly. In this study, we use the comprehensive geriatric assessment to study the effects of surgery and anesthesia on elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participants receiving general anesthesia for longer than 1 hour.

Exclusion Criteria:

* Participants receiving local anesthesia.
* Participants receiving regional anesthesia.
* Participants receiving general anesthesia for less than 1 hour.
* Participants with psychiatric disorder.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The elderly population requiring anesthesia.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental Status Examination | Before general anesthesia till 48-hours post-anesthesia.
  The Mini-Mental Status Examination is a screening tool for dementia. The investigator asks the patient a series of questions to which the patient answers to his or her best ability.
  Minium score of zero and a maximum score of 30. Lower value represents a worse outcome.
  A score of less than 24 is considered abnormal.
Geriatric Depression Scale - 15 | Before general anesthesia till 48-hours post-anesthesia.
  The Geriatric Depression Scale (short form) is a screening tool for depression. It is a questionnaire composed of 15 questions. The investigator asks the patient 15 questions in which the patient answers "yes" or "no".
  Each question weighs 1 point with a minimum score of zero and maximum score of 15.
  The higher the score, the more likely depression is present. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
Confusion Assessment Method | Before general anesthesia till 48-hours post-anesthesia.
  The Confusion Assessment Method is a screening tool for delirium. It comprises of four parts: "(1) acute onset and fluctuating course", "(2) inattention", "(3) disorganized thinking", and "(4) altered level of consciousness".
  "(1) Acute onset and fluctuating course" has two questions and the rest with one question each.
  The investigator conducts the assessment with the patient answering "yes" or "no" to each question.
  Delirium is diagnosed under these scenarios: yes to all four questions, yes to (1)+(2)+(3), yes to (1)+(2)+(4).
Barthel Index | Before general anesthesia till 48-hours post-anesthesia.
  Barthel Index is an ordinal scale used to measure performance in ADL (activities of daily living).
  It comprises of ten variables describing ADL. A minium of zero and a maximum and 100 is scored. Higher score reflects greater ability to function independently. 60 or less is classified as dependent. Scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan